CLINICAL TRIAL: NCT06510413
Title: An Bioequivalence Study of Loxoprofen Sodium Patches in Chinese Healthy Volunteers
Brief Title: An Bioequivalence Study of Loxoprofen Sodium Patches in Healthy Volunteers
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Frontier Biotechnologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: JY-BE-LSLF-2024-042
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Osteoarthritis; Muscle Pain; Swelling Muscle
MeSH Terms: conditions — Osteoarthritis; Myalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Loxoprofen Sodium Patches (Sequence TR) (Other): Dosage form: patch
  Dosage: 100 mg/ patch
  Frequency and duration: single dose
  Subjects receive the test product (T) in the first period, then the reference product (R) in the second period.
  Interventions: Drug: Loxoprofen Sodium Patches(reference product); Drug: Loxoprofen Sodium Patches(test product )
- Loxoprofen Sodium Patches (Sequence RT) (Other): Dosage form: patch
  Dosage: 100 mg/ patch
  Frequency and duration: single dose
  Subjects receive the reference product (R) in the first period, then the test product (T) in the second period
  Interventions: Drug: Loxoprofen Sodium Patches(reference product); Drug: Loxoprofen Sodium Patches(test product )

INTERVENTIONS:
Drug: Loxoprofen Sodium Patches(reference product) — Single dose of one patch in each period; Apply for 24 hours each time
  Other Names: Loxonin®
Drug: Loxoprofen Sodium Patches(test product ) — Single dose of one patch in each period; Apply for 24 hours each time
  Other Names: FB3002

SUMMARY:
This study was a single-center, randomized, open-label, two-agent, two-cycle, double-cross bioequivalence trial.

DETAILED DESCRIPTION:
The objectives of this study are to evaluate the difference of absorption degree and absorption rate of two kinds of patches( FB3002 vs. Loxonin®) in Chinese healthy population, and to assess the bioavailability of these two patches.

ELIGIBILITY:
Inclusion Criteria:

* Male weight ≥50 kg, female weight ≥45 kg, body mass index (BMI) between 19.0 and 28.0 kg/m2, inclusive .
* Informed consent: signed written informed consent before inclusion in the study.
* The subjects are well communicated and are able to comply with the requirements of the study

Exclusion Criteria:

* Participated in other drug intervention studies within 90 days
* Allergic to this product and excipients, or have a history of food, drug allergy or other allergic diseases (asthma, urticaria, eczema dermatitis, etc.)
* Aspirin asthma
* Any visible skin disorder or abnormal skin pigmentation which, in the opinion of the investigator, would interfere with the outcome of the trial.
* A history of cardiovascular system, respiratory system, digestive system, urinary system, endocrine system, immune system, nervous/psychiatric system, blood and lymphatic system, and skeletal musculoskeletal system that investigator have determined to be abnormal and clinically significant
* Postural hypotension, needle fainting or blood fainting history or venipuncture intolerance
* Any drug that inhibits or induces liver metabolism has been used in the 30 days prior to screening. Inducers: barbiturates, carbamazepine, phenytoin sodium, glucocorticoids, omeprazole; Inhibitors: SSRI antidepressants, cimetidine, Diltiazem, nitroimidazoles, sedatives and hypnotics, verapamil, fluoroquinolones, antihistamines
* Blood donation or significant blood loss (>400 mL, except for female menstrual period) in the 3 months prior to screening, blood transfusion or use of blood products, or have a blood donation plan during/within 3 months after the study
* Smoked more than 5 cigarettes per day in the 3 months prior to screening, or unwilling to prohibit the use of any tobacco products during the trial period
* History of alcohol abuse within 6 months
* Subjects who consumed excessive amounts of tea, coffee or caffeinated beverages within 3 months, or who did not agree to the prohibition of tea, coffee or caffeinated beverages in the study
* Subjects who have special requirements for diet and cannot comply with a unified diet
* History of drug abuse within 1 year
* Subjects who have unprotected sex in 2 weeks, or planned to have a child during the study period, planned to donate sperm and eggs, or are unwilling to use one or more non-drug contraceptive methods during the study, or are unwilling to use contraception within 3 months after the study
* Pregnant or nursing women
* Positive skin scratch test positive
* Clinically significant vital signs laboratory, physical examination, or 12-lead electrocardiogram abnormalities as judged by the investigator
* Other situations that the investigator determines are not suitable for participating in this clinical trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Cmax of loxoprofen and its trans-OH | 0-72 hours
  Maximum plasma concentration. Analyzing AUC with ANOVA test to evaluate the 90% confidence interval for the ratio (Test/Reference) of the population mean with a logarithmic transformation prior to analysis with acceptance interval of 0.80 - 1.25.
AUC0-T of loxoprofen and its trans-OH | 0-72 hours
  Area under the plasma concentration curve from time 0 to the last measured (AUC0-t).
  Analyzing AUC with ANOVA test to evaluate the 90% confidence interval for the ratio (Test/Reference) of the population mean with a logarithmic transformation prior to analysis with acceptance interval of 0.80 - 1.25.
AUC0-∞ of loxoprofen and its trans-OH | 0-72 hours
  Area under the plasma concentration curve from time 0 to ∞ (AUC0-∞). Analyzing AUC with ANOVA test to evaluate the 90% confidence interval for the ratio (Test/Reference) of the population mean with a logarithmic transformation prior to analysis with acceptance interval of 0.80 - 1.25.

SECONDARY OUTCOMES:
Adverse Events | 0-14 days
  All of the adverse events will be reported
Tmax of loxoprofen and its trans-OH | 0-72 hours
  Time to reach maximum plasma concentration
t1/2 of loxoprofen and its trans-OH | 0-72 hours
  Apparent terminal elimination half-life
λz | 0-72 hours
  Apparent terminal elimination rate constant
AUC_%Extrap | 0-72 hours
  Percentage of AUCINF(_obs, _pred) due to extrapolation from Tlast to infinity
Irritation score | 0-14 days
  A combined irritation score should be calculated by adding the "dermal response" score and the numeric equivalent for "other effects" letter score.

CONTACTS AND LOCATIONS:
Overall Officials: Cheng Yao, Study Director — Frontier Biotechnologies Inc.